CLINICAL TRIAL: NCT00839111
Title: A Phase Ⅱ Open Label, Non Randomized Study, in Which Sorafenib is Used in Combination With Irinotecan, Leucovorin and Fluorouracil in Patients With Advanced Colorectal Cancer After Failure of Oxaliplatin Treatment
Brief Title: Sorafenib and FOLFIRI Regimen in 2nd Colorectal Cancer (CRC) After Failure of Oxaliplatin Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Base for drug clinical trials, Fudan University,cancer hospital., Department of Medical Oncology, Cancer Hospital, Fuandan University.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bay43-9006-2008005
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2010-09-15 (Estimated); Status verified 2010-09

CONDITIONS: Colorectal Neoplasms
Keywords: Progression free survival; Toxicity; Response rate; overall survival
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Sorafenib; IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Sorafenib plus FOLFIRI regimen
  Interventions: Drug: sorafenib; Drug: FOLFIRI

INTERVENTIONS:
Drug: sorafenib — Sorafenib 400mg twice daily from d3 to d14,d17-28
  Other Names: Nexavar
Drug: FOLFIRI — Irinotecan 180 mg/m2,CF 400mg/m2 5Fu 400mg/m2 bolus, followed by 2.4g/m2 continuously intravenous infusion for 46 hours, days 1 and 15, every 4 weeks per cycle
  Other Names: Irinotecan:Campto

SUMMARY:
The purpose of this study is to evaluate the Progression-Free Survival (PFS) time of Sorafenib in combination with FOLFIRI regimen used as in the second front treatment in patients with advanced CRC after failure of oxaliplatin treatment.

DETAILED DESCRIPTION:
This is a phase Ⅱ open label, non randomized study, in which sorafenib is used in combination with irinotecan, leucovorin and fluorouracil in patients with advanced colorectal cancer after failure of oxaliplatin treatment.The aim of this study is to determine the Progression-Free Survival (PFS) of Sorafenib used in combination with FOLFIRI regimen as a second front treatment in patients with advanced CRC after failure of oxaliplatin treatment, defined as the time from treatment to disease progression or death due to any cause. The other secondary endpoints are disease control rate, defined as complete response, partial response, and stable disease.Response rate,overall survival, and safety are also evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent
2. Histological or cytological confirmed adenocarcinoma of the colon or rectum
3. Age between 18 and 75 years.
4. Patient with metastatic disease failed after at least 2 cycles of oxaliplatin-based systemic chemotherapy, excluding adjuvant chemotherapy. Disease progression should be proven by radiological evidence. A duration of 28 days after oxaliplatin therapy is also required.
5. ECOG Performance Status of 0 or1
6. Life expectancy of at least 12 weeks
7. The required evidence of measurable lesions should be at least 10 mm in the longest diameter by spiral computed tomography scan or 20 mm with conventional techniques (RECIST criteria)
8. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:

   * Hemoglobin > 9.0 g/dl
   * Absolute neutrophil count (ANC) >1,500/mm3
   * Platelet count 100,000/μl
   * Total bilirubin < 1.5 times the upper limit of normal ALT and AST < 2.5 x ULN(< 5 x ULN for patients with liver involvement of their cancer)
   * ALP< 4 x ULN
   * PT-INR/PTT < 1.5 x upper limit of normal
   * Serum creatinine < 1.5 x ULN

Exclusion Criteria:

1. Patients unable to swallow oral medications
2. History of cardiac disease:

   * congestive heart failure >NYHA class 2
   * active CAD (MI more than 6 mo prior to study entry is allowed)
   * cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted) or uncontrolled hypertension
3. History of HIV infection or chronic hepatitis B or C (high copy number of HBV).
4. Active clinically serious infections (> grade 2 NCI-CTC version 3.0)
5. Symptomatic metastatic brain or meningeal tumors (unless the patient is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry)
6. Patients with seizure disorder requiring medication (such as steroids or anti-epileptics)
7. History of organ allograft ,The organ allograft may be allowed as protocol specific.
8. Patients undergoing renal dialysis
9. Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma within 5 years.
10. Patients with evidence or history of bleeding diathesis.Significant haemorrhage (>30 ml/bleeding episode in previous 3 months),haemoptysis (>5 ml fresh blood in previous 4 weeks) or thrombotic event (including transient ischaemic attack) in the previous 12 months.
11. chronic inflammatory bowel disease; ileus; genetic fructose intolerance
12. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
13. Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study
14. Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial (and men for at least 3 months after last administration of study medication).
15. Prior exposure to the study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-11 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) ,defined as the time from treatment to disease progression or death due to any cause | every 8 weeks

SECONDARY OUTCOMES:
Secondary endpoints are disease control rate, defined as a complete response, partial response, and stable disease; Response rate and overall survival; and safety are also evaluated. | every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, MD, Principal Investigator — Cancer Hospital,Fudan University
Locations (1):
- Cancer Hospital,Fudan University, Shanghai, Shanghai Municipality, China